CLINICAL TRIAL: NCT00035555
Title: Phase II/III, Open-Label, Randomized, Controlled, Multiple-Dose Study of Efficacy and Safety of BMS-224818 (Belatacept) as Part of a Quadruple Drug Regimen in First Renal Transplant Recipients
Brief Title: Study Comparing the Safety and Efficacy of Belatacept With That of Cyclosporine in Patients With a Transplanted Kidney
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IM103-100
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-11

CONDITIONS: Graft Rejection; Kidney Transplantation; Renal Transplantation
Keywords: kidney; transplant; rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Abatacept; Cyclosporine; Mycophenolic Acid; Adrenal Cortex Hormones

ARMS (3):
- Belatacept: More intensive (MI) regimen (Experimental): The MI regimen was designed to achieve projected serum trough concentrations of belatacept of approximately 20 μg/mL through Day 99, and approximately 5 μg/mL through Day 183 (10 mg/kg on Days 1, 5, 15, 29, 43, 57, 71, 85, 113, 141, and 169). After Day 169, patients were reallocated and dosed to achieve projected trough serum concentrations of approximately 2 or 0.25 μg/mL (5 mg/kg every 4 or 8 weeks starting on Day 197). Those patients who received belatacept every 8 weeks received placebo infusions on scheduled treatment dates between infusions of active drug to maintain the blind between treatment regimens. Patients initially received mycophenolate mofetil (MMF), 2 g/d orally, unless the investigator chose to administer ≥1 doses intravenously The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the patient was able to tolerate medications by mouth. Corticosteroids given daily.
  Interventions: Drug: Belatacept; Drug: Mycophenolate mofetil (MMF); Drug: Corticosteroids
- Belatacept: Less intensive (LI) regimen (Experimental): The LI regimen was designed to achieve projected trough serum concentrations of belatacept of approximately 20 μg/mL through Day 29, and approximately 5 μg/mL through Day 99 (10 mg/kg on Days 1, 15, 29, 57 and 85). After Day 85, these subjects were reallocated and dosed to achieve projected trough serum concentrations of either approximately 2 or 0.25 μg/mL (5 mg/kg every 4 or 8 weeks starting on Day 113). Participants initially received mycophenolate mofetil (MMF), 2 g/d orally, unless the investigator chose to administer ≥1 doses intravenously The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. Corticosteroids given daily.
  Interventions: Drug: Belatacept; Drug: Mycophenolate mofetil (MMF); Drug: Corticosteroids
- Cyclosporine regimen (Experimental): The initial daily dose was 7±3 mg/kg. Subsequent doses were adjusted to maintain a predefined range of serum concentrations: 1st month, target level 150-400 ng/mL; after 1st month, target level of 150-300 ng/mL. Participants initially received mycophenolate mofetil (MMF), 2 g/d orally, unless the investigator chose to administer ≥1 doses intravenously The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. Corticosteroids given daily.
  Interventions: Drug: Cyclosporine; Drug: Mycophenolate mofetil (MMF); Drug: Corticosteroids

INTERVENTIONS:
Drug: Belatacept — Solution, intravenous
  Other Names: LEA29Y, BMS-224818
  Arms: Belatacept: Less intensive (LI) regimen; Belatacept: More intensive (MI) regimen
Drug: Cyclosporine — Oral, capsule
  Other Names: The cyclosporine used in this study will be in the modified formulation with enhanced bioavailability.
  Arms: Cyclosporine regimen
Drug: Mycophenolate mofetil (MMF) — Oral, capsule
Drug: Corticosteroids — Corticosteroids given daily, orally or intravenously (IV). Day of transplant (Day 1): methylprednisolone, 500 mg, given IV on arrival in operating room; Day 2: methylprednisolone, 250 mg, given IV once daily; Day 3: prednisone, 100 mg, given orally once daily; Day 4: prednisone, 50 mg, given orally once daily; Days 5 through 30: prednisone, 25 mg, given orally once daily; Days 31-44: prednisone, 22.5 mg, given orally once daily; Days 45-58: prednisone, 20 mg, given orally once daily

SUMMARY:
The purpose of this study is to determine whether treatment with Belatacept (BMS-224818) is as efficacious as treatment with cyclosporine at preventing acute rejection and with a superior safety/tolerability profile (better kidney function and blood pressure, fewer lipid problems, less diabetes mellitus).

ELIGIBILITY:
Key inclusion criteria

* Recipients of first kidney transplant

Key exclusion criteria

* Those at high risk for acute allograft rejection, including those who receive a second or more renal transplant, those with a history of panel reactive antibody levels >20%, and those considered by investigators to be at relatively higher risk for acute rejection
* Human leukocyte antigen-identical donor-recipient pairs
* Cold ischemia time >36 hours (donor kidney)
* Participants who are positive for hepatitis C antibody, on polymerase chain reaction, for hepatitis B surface antigen, and for human immunodeficiency virus
* A positive purified protein derivative tuberculosis test (test performed within 1 year of enrollment), unless previously vaccinated with Bacille-Calmette-Guérin or those who had a history of adequate chemoprophylaxis
* Any active infection that would normally exclude transplantation
* Recipients of multiple organ transplants
* Donor age >60 or <6 years or donors whose hearts were not beating
* Recipients with underlying renal disease of (due to risk of rapid disease recurrence in the allograft): focal segmental glomerulosclerosis, Type I or II membranoproliferative glomerulonephritis, or hemolytic uremic syndrome/ thrombotic thrombocytopenic purpura
* A positive T-cell lymphocytoxic crossmatch using donor lymphocytes and recipient serum
* A history of true allergy to intravenous iodinated roentgenographic contrast agents
* Participants with life expectancy severely limited by disease state or other underlying medical condition
* A history of cancer (other than nonmelanoma skin cell cancers cured by local resection) within the last 5 years
* Mammogram film with any clinically significant abnormality requiring further investigation or biopsies
* History of substance abuse (drug or alcohol) or psychotic disorders that were not compatible with adequate study follow-up
* A currently functioning, nonrenal transplant
* Previous treatment with basiliximab for any reason
* Active peptic ulcer disease, chronic diarrhea, or gastrointestinal malabsorption
* Those who had used any investigational drug within 30 days before the Day 1 visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2001-03; Primary Completion 2004-01 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Univ. of Calif. - San Francisco, San Francisco, California
  - Emory Univ. School of Medicine, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Univ. of Nebraska Medical Center, Omaha, Nebraska
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Univ. of Pennsylvania, Philadelphia, Pennsylvania
  - Medical Univ. of South Carolina, Charleston, South Carolina
  - Baylor Univ. Medical Center, Dallas, Texas
  - Univ. of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 230 participants who had undergone transplantation were enrolled
Groups:
- Belatacept: More Intensive (MI) Regimen: The MI regimen aimed to achieve projected serum trough concentrations of belatacept of 20 μg/mL through Day 99, and 5 μg/mL through Day 183 (10 mg/kg on Days 1, 5, 15, 29, 43, 57, 71, 85, 113, 141 and 169). After Day 169, doses were reassigned to achieve projected trough serum concentrations of 2 or 0.25 μg/mL (5 mg/kg every 4 or 8 weeks starting on Day 197). Participants initially received mycophenolate mofetil (MMF), 2 g/d orally or ≥1 doses intravenously (IV),depending on the investigators decision. The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. All participants also received induction therapy (2 doses) with basiliximab IV and daily corticosteroids.
- Belatacept: Less Intensive (LI) Regimen: The LI regimen was designed to achieve projected trough serum concentrations of belatacept of 20 μg/mL through Day 29, and approximately 5 μg/mL through Day 99 (10 mg/kg on Days 1, 15, 29, 57 and 85). After Day 85, these subjects were reallocated and dosed to achieve projected trough serum concentrations of either 2 or 0.25 μg/mL (5 mg/kg every 4 or 8 weeks starting on Day 113). Participants initially received mycophenolate mofetil (MMF), 2 g/d orally or ≥1 doses intravenously (IV),depending on the investigators decision. The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. All participants also received induction therapy (2 doses) with basiliximab IV and daily corticosteroids.
- Cyclosporine Regimen: Cyclosporine regimen was designed to achieve a specified range of target serum concentrations consistent with current medical practice for the duration of the study. The initial daily dose was 7±3 mg/kg. Subsequent doses were adjusted to maintain a predefined range of serum concentrations: 1st month, target level 150-400 ng/mL; after 1st month, target level of 150-300 ng/mL. Participants initially received mycophenolate mofetil (MMF), 2 g/d orally or ≥1 doses intravenously (IV),depending on the investigators decision. The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. All participants also received induction therapy (2 doses) with basiliximab IV and daily corticosteroids.
Period: Overall Study
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Started | 74 (Randomized patients) | 71 (Randomized patients) | 73 (Randomized patients)
Number Who Had Undergone Transplantation | 74 | 71 | 73
Number Who Received Study Drug | 74 | 71 | 71
Completed | 58 | 55 | 51
Not Completed | 16 | 16 | 22
Not completed — Adverse Event | 5 | 8 | 9
Not completed — Allograft loss | 1 | 1 | 2
Not completed — Death | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Noncompliance | 0 | 1 | 1
Not completed — Prohibited medication | 1 | 1 | 0
Not completed — Treatment failure/lack of efficacy | 7 | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Investigator deemed not a good candidate | 0 | 0 | 1
Not completed — Received cyclosporin in error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for all patients who were randomized and received transplants; participant flow is provided for all randomized participants who received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen | Total
Number analyzed (Participants) | 74 | 71 | 73 | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (10.8) | 42.1 (11.6) | 46.1 (10.9) | 44.9 (11.2)
Age, Continuous [Median (Full Range); unit: Years] | 45.5 [23.0 to 70.0] | 43.0 [18.0 to 71.0] | 46.0 [23.0 to 66.0] | 45.0 [18.0 to 71.0]
Age, Customized [Number; unit: Participants]
  Between 18 and 45 years | 37 | 42 | 36 | 115
  Between 46 and 60 years | 31 | 26 | 33 | 90
  Older than 60 years | 6 | 3 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 24 | 67
  Male | 54 | 48 | 49 | 151
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 64 | 57 | 59 | 180
  Black or African American | 6 | 6 | 6 | 18
  Asian/Pacific Islander | 3 | 4 | 5 | 12
  Hispanic | 1 | 4 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Episode of Clinically-suspected and Biopsy-proven Acute Rejection (CSPAR)
Description: No participant was to receive treatment for acute rejection without a biopsy to confirm the diagnosis. CSPAR=Clinically-suspected rejection, defined as an increase in serum creatinine ≥0.5 mg/dL compared with the baseline value in the absence of other factors known to adversely affect renal function, and biopsy-proven rejection, which includes all cases in which a biopsy was read by the central pathologist as demonstrating acute rejection regardless of the reason why the biopsy was performed.
Time Frame: By Month 6 posttransplant (From Day 1 to Month 6)
Population: All randomized participants who underwent transplantation
Measure: Number; unit: Participants
Groups:
- Cyclosporine Regimen: The cyclosporine regimen was designed to achieve a specified range of target serum concentrations consistent with current medical practice for the duration of the study. The initial daily dose was 7±3 mg/kg. Subsequent doses were adjusted to maintain a predefined range of serum concentrations: 1st month, target level 150-400 ng/mL; after 1st month, target level of 150-300 ng/mL. Participants initially received mycophenolate mofetil (MMF), 2 g/d orally or ≥1 doses intravenously (IV),depending on the investigators decision. The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. All participants also received induction therapy (2 doses) with basiliximab IV and daily corticosteroids.
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
Participants | 5 [1.0 to 12.5] | 4 | 6

2. Secondary Outcome: Percentage of Participants With Biopsy-proven Acute Rejection (BPAR) Through Months 6 and 12
Description: BPAR includes all cases in which a biopsy read by the central pathologist demonstrates acute rejection, regardless of the reason that the biopsy was performed.
Time Frame: Through Months 6 and 12 posttransplant (From Day 1 to Months 6 and 12)
Population: All randomized participants who underwent transplantation
Measure: Number; unit: Percentage of participants
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
Percentage of participants
  Up to 6 months | 14.9 | 23.9 | 17.8
  Up to 12 months | 18.9 | 29.6 | 17.8

3. Secondary Outcome: Percentage of Participants With Biopsy-proven Acute Rejection (BPAR) or Who Received Treatment for Acute Rejection
Description: BPAR includes all cases in which a biopsy read by the central pathologist demonstrates acute rejection, regardless of the reason that the biopsy was performed. A participant was reported as having had an episode of treated acute rejection if he or she received antirejection therapy during an episode of rejection (clinically-suspected or biopsy-proven rejection).
Time Frame: By Months 3, 6, and 12 posttransplant (Day 1 to Months 3, 6, and 12)
Population: All randomized participants who underwent transplantation
Measure: Number; unit: Percentage of participants
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
Percentage of participants
  By Month 3 | 21.6 | 29.6 | 17.8
  By Month 6 | 23.0 | 32.4 | 24.7
  By Month 12 | 28.4 | 38.0 | 27.4

4. Secondary Outcome: Percentage of Participants With Acute Rejection or Presumed Acute Rejection (PAR)
Description: Throughout this study, acute rejection=clinically-suspected and biopsy-proven acute rejection (BPAR). Clinically-suspected rejection is defined as an increase in serum creatinine ≥0.5 mg/dL compared with the baseline value in the absence of other factors known to adversely affect renal function. BPAR includes all cases in which a biopsy was read by the central pathologist as demonstrating acute rejection regardless of the reason why the biopsy was performed. PAR is defined as an elevation in SCr ≥0.5 mg/dL compared with the baseline value in the absence of other factors known to adversely affect renal function that led the investigator to suspect that the participant had experienced acute rejection, and in whom either the biopsy did not confirm acute rejection and the participant received treatment for acute rejection or the participant received treatment for acute rejection without a biopsy to confirm the diagnosis.
Time Frame: By Months 6 and 12 posttransplant (Day 1 to Months 6 and 12)
Population: All randomized participants who underwent transplantation
Measure: Number; unit: Percentage of participants
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
Percentage of participants
  Month 6: Acute rejection or PAR | 11 | 9 | 10
  Month 12: Acute rejection or PAR | 11 | 10 | 11
  Month 6: PAR | 5 | 3 | 1
  Month 12: PAR | 5 | 4 | 3

5. Secondary Outcome: Percentage of Participants Who Had Chronic Allograft Nephropathy
Description: Based on postbaseline biopsies
Time Frame: By Months 6 and 12 posttransplant (Day 1 to Months 6 and 12)
Population: All randomized participants who underwent transplantation and who had at least 1 biopsy following Day 1; n=evaluable participants
Measure: Number; unit: Percentage of participants
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
Percentage of participants
  Month 6 (n= 32, 33, 27) | 18.8 | 9.1 | 33.3
  Month 12 (n=52, 54, 45) | 28.8 | 20.4 | 44.4

6. Secondary Outcome: Mean Iohexol Clearance
Description: Iohexol, a true glomerular filtration marker, is used to measure glomerular filtration rate.
Time Frame: By Months 1, 6, and 12 posttransplant (Day 1 to Months 1, 6, and 12)
Population: All randomized participants who underwent transplantation
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
mL/min per 1.73 m^2
  Month 1 (n=53, 51, 48) | 59.7 (17.3) | 60.2 (14.4) | 54.0 (19.3)
  Month 6 (n=41, 41, 31) | 62.2 (25.6) | 64.5 (19.5) | 56.0 (19.5)
  Month 12 (n=32, 37, 27) | 66.3 (20.7) | 62.1 (15.9) | 53.5 (16.4)

7. Secondary Outcome: Percentage of Participants Who Used Antihypertensive Medication
Description: Hypertension is defined as diastolic blood pressure ≥90 mm Hg and/or systolic blood pressure ≥140 mm Hg
Time Frame: By Months 6 and 12 posttransplant (Day 1 to Months 6 and 12)
Population: All randomized participants who underwent transplantation
Measure: Number; unit: Percentage of participants
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
Percentage of participants
  Month 6: Total requiring at least 1 medication | 87.7 | 78.6 | 88.4
  Month 6: Requiring 1 medication | 24.7 | 27.1 | 21.7
  Month 6: Requiring 2 medications | 23.3 | 28.6 | 31.9
  Month 6: Requiring 3 medications | 23.3 | 14.3 | 21.7
  Month 6: Requiring 4 medications | 11.0 | 7.1 | 11.6
  Month 6: Requiring 5 medications | 2.7 | 1.4 | 1.4
  Month 6: Requiring 6 medications | 2.7 | 0.0 | 0.0
  Month 6: Requiring >6 medications | 0.0 | 0.0 | 0.0
  Month 12: Total requiring at least 1 medication | 79.7 | 71.6 | 86.4
  Month 12: Requiring 1 medication | 21.7 | 26.9 | 20.3
  Month 12: Requiring 2 medications | 23.2 | 9.0 | 22.0
  Month 12: Requiring 3 medications | 23.2 | 9.0 | 22.0
  Month 12: Requiring 4 medications | 8.7 | 7.5 | 15.3
  Month 12: Requiring 5 medications | 5.8 | 0.0 | 3.4
  Month 12: Requiring 6 medications | 1.4 | 0.0 | 0.0
  Month 12: Requiring >6 medications | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Number of Participants With Hypertension
Description: Hypertension is defined as diastolic blood pressure ≥90 mm Hg and/or systolic blood pressure ≥140 mm Hg or, the use of any antihypertensive medication.
Time Frame: By Months 6 and 12 posttransplant (Day 1 to Months 6 and 12)
Population: All randomized participants who underwent transplantation
Measure: Number; unit: Participants
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
Participants
  At Month 6 | 16 | 15 | 18
  At Month 12 | 14 | 12 | 11

9. Other Pre Specified Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, Discontinuations Due to SAEs, Adverse Events (AEs), Treatment-related AEs, and Discontinuations Due to AEs
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Day 1 (posttransplant) continuously to 56 days following last dose of study medication
Population: All randomized participants who underwent transplantation and who received treatment
Measure: Number; unit: Participants
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 71
Participants
  Deaths | 0 | 0 | 2
  SAEs | 50 | 52 | 42
  Treatment-related SAEs | 21 | 23 | 21
  Discontinuations due to SAEs | 13 | 14 | 10
  AEs | 73 | 69 | 68
  Treatment-related AEs | 43 | 40 | 50
  Discontinuations due to AEs | 13 | 15 | 14

10. Secondary Outcome: Mean LDL Cholesterol, HDL Cholesterol, Total Cholesterol, Triglyceride, and Non-HDL Levels
Description: LDL=low-density lipoprotein; HDL=high-density lipoprotein. Total cholesterol=LDL + HDL + very low-density (VLDL) cholesterol. VLDL=triglycerides divided by 5. Non-HDL cholesterol=Total cholesterol minus HDL cholesterol.
Time Frame: By Months 1, 6, and 12 posttransplant (Day 1 to Months 1, 6, and 12)
Population: All randomized participants who received a transplant; n=evaluable participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 74 | 71 | 73
mg/dL
  LDL cholesterol: Month 1 (n=69, 69, 66) | 129 (48.9) | 120 (33.2) | 137 (42.9)
  LDL cholesterol: Month 6 (n=63, 66, 55) | 125 (33.9) | 121 (39.2) | 131 (41.4)
  LDL cholesterol: Month 12 (n=61, 60, 52) | 120 (33.8) | 125 (32.0) | 125 (36.4)
  HDL cholesterol: Month 1 (n=68, 68, 64) | 64 (19.4) | 68 (21.7) | 70 (21.6)
  HDL cholesterol: Month 6 (n=62, 65, 62) | 54 (14.8) | 56 (19.0) | 62 (20.1)
  HDL cholesterol: Month 12 (n=60, 57, 48) | 53 (15.7) | 56 (13.5) | 59 (18.5)
  Total cholesterol: Month 1 (n=69, 69, 65) | 222 (64.7) | 210 (45.6) | 239 (53.7)
  Total cholesterol: Month 6 (n=63, 65, 54) | 204 (40.4) | 202 (47.7) | 224 (54.8)
  Total cholesterol: Month 12 (n=60, 58, 50) | 198 (41.4) | 201 (40.0) | 212 (44.2)
  Triglycerides: Month 1 (n=69, 69, 65) | 168 (125.3) | 147 (65.3) | 185 (103.9)
  Triglycerides: Month 6 (n=63, 65, 54) | 177 (113.1) | 168 (87.4) | 198 (119.7)
  Triglycerides: Month 12 (n=60, 58, 50) | 176 (87.9) | 152 (63.5) | 186 (91.6)
  Non-HDL: Month 1 (n=68, 68, 64) | 159 (62.7) | 142 (40.2) | 169 (51.5)
  Non-HDL cholesterol: Month 6 (n=62, 64, 51) | 150 (39.4) | 143 (42.1) | 165 (55.1)
  Non-HDL cholesterol: Month 12 (n=59, 56, 48) | 145 (36.7) | 144 (35.8) | 151 (43.4)

11. Secondary Outcome: Number of Participants With Posttransplant Diabetes Mellitus
Description: Posttransplant diabetes mellitus is defined as the need for treatment of hyperglycemia with either an oral agent or insulin for a total of >4 weeks or hemoglobin A1c (HbA1c) >7% in a participant not known to be diabetic prior to transplantation
Time Frame: By Months 1, 3, 6, 9, and 12 posttransplant (Day 1 to Months 1, 3, 6, 9, and 12 )
Population: All randomized participants who received transplants and who were not known to be diabetic prior to transplant
Measure: Number; unit: Participants
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept: Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 67 | 65 | 60
Participants
  Up to Month 1: All events | 5 | 0 | 1
  Month 1: Hyperglycemia medication | 0 | 0 | 1
  Month 1: HbA1c >7% | 5 | 0 | 0
  Up to Month 3: All events | 5 | 1 | 3
  Up to Month 3: Hypoglycemic medication | 0 | 0 | 2
  Up to Month 3: HbA1c >7% | 5 | 1 | 1
  Up to Month 6: All events | 6 | 3 | 4
  Up to Month 6: Hyperglycemia medication | 0 | 0 | 2
  Up to Month 6: HbA1c >7% | 6 | 3 | 2
  Up to Month 9: All events | 8 | 3 | 5
  Up to Month 9: Hyperglycemia medication | 2 | 0 | 2
  Up to Month 9: HbA1c >7% | 7 | 3 | 3
  Up to Month 12: All events | 8 | 4 | 7
  Up to Month 12: Hyperglycemia medication | 2 | 0 | 3
  Up to Month 12: HbA1c >7% | 7 | 4 | 4

12. Other Pre Specified Outcome: Number of Participants Meeting Marked Abnormality Criteria for Select Hemolytic, Blood Chemistry, and Urinalysis Laboratory Test Results
Description: Normal laboratory values: Hemoglobin (g/dL): Males (18-64 years) 13.8-17, (65 years and older) 11.8-16.8; Females (18-64 years) 12.0-15.6, F (65 years and older) 11.1-15.5. Platelets (per mm^3) 130,000-400,000. Leukocytes (18 years and older) 3.8-10.8 1000/uL. ALT (u/L)(13 years and older) 0-48.
Time Frame: Days 8 and Months 1, 3, 6, 9, and 12 posttransplant (from Day 1)
Population: All randomized participants who underwent transplantation and who received treatment
Measure: Number; unit: Participants
Groups:
- Belatacept:Less Intensive (LI) Regimen: The LI regimen was designed to achieve projected trough serum concentrations of belatacept of 20 μg/mL through Day 29, and approximately 5 μg/mL through Day 99 (10 mg/kg on Days 1, 15, 29, 57 and 85). After Day 85, these subjects were reallocated and dosed to achieve projected trough serum concentrations of either 2 or 0.25 μg/mL (5 mg/kg every 4 or 8 weeks starting on Day 113). Participants initially received mycophenolate mofetil (MMF), 2 g/d orally or ≥1 doses intravenously (IV),depending on the investigators decision. The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. All participants also received induction therapy (2 doses) with basiliximab IV and daily corticosteroids.
Arm/Group | Belatacept: More Intensive (MI) Regimen | Belatacept:Less Intensive (LI) Regimen | Cyclosporine Regimen
Number analyzed (Participants) | 72 | 70 | 69
Participants
  Hemoglobin, low | 13 | 7 | 9
  Hemoglobin, high | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Platelet count, low | 1 | 0 | 3
  Platelet count, high | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Leukocytes, low | 1 | 4 | 5
  Leukocytes, high | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Alanine aminotransferase (ALT), low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  ALT, high | 9 | 3 | 7

ADVERSE EVENTS:
Description: Includes all randomized participants who underwent transplantation and received treatment
Groups:
- Belatacept: Less-intensive (LI) Regimen: The LI regimen was designed to achieve projected trough serum concentrations of belatacept of 20 μg/mL through Day 29, and approximately 5 μg/mL through Day 99 (10 mg/kg on Days 1, 15, 29, 57 and 85). After Day 85, these subjects were reallocated and dosed to achieve projected trough serum concentrations of either 2 or 0.25 μg/mL (5 mg/kg every 4 or 8 weeks starting on Day 113). Participants initially received mycophenolate mofetil (MMF), 2 g/d orally or ≥1 doses intravenously (IV),depending on the investigators decision. The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. All participants also received induction therapy (2 doses) with basiliximab IV and daily corticosteroids.
- Belatacept: More-intensive (MI) Regimen: The MI regimen aimed to achieve projected serum trough concentrations of belatacept of 20 μg/mL through Day 99, and 5 μg/mL through Day 183 (10 mg/kg on Days 1, 5, 15, 29, 43, 57, 71, 85, 113, 141 and 169). After Day 169, doses were reassigned to achieve projected trough serum concentrations of 2 or 0.25 μg/mL (5 mg/kg every 4 or 8 weeks starting on Day 197). Participants initially received mycophenolate mofetil (MMF), 2 g/d orally or ≥1 doses intravenously (IV),depending on the investigators decision. The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. All participants also received induction therapy (2 doses) with basiliximab IV and daily corticosteroids.
- Cyclosporin Regimen: The cyclosporine regimen was designed to achieve a specified range of target serum concentrations consistent with current medical practice for the duration of the study. The initial daily dose was 7±3 mg/kg. Subsequent doses were adjusted to maintain a predefined range of serum concentrations: 1st month, target level 150-400 ng/mL; after 1st month, target level of 150-300 ng/mL. Participants initially received mycophenolate mofetil (MMF), 2 g/d orally or ≥1 doses intravenously (IV),depending on the investigators decision. The first MMF dose was administered preoperatively; subsequent doses were administered in 2 or 3 divided doses, every 8-12 hours, beginning as soon as the participant was able to tolerate medications by mouth. All participants also received induction therapy (2 doses) with basiliximab IV and daily corticosteroids.
Arm/Group | Belatacept: Less-intensive (LI) Regimen | Belatacept: More-intensive (MI) Regimen | Cyclosporin Regimen
Serious Adverse Events (participants affected / at risk) | 52/71 | 50/74 | 42/71
Other Adverse Events (participants affected / at risk) | 66/71 | 68/74 | 67/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept: Less-intensive (LI) Regimen (N=71) | Belatacept: More-intensive (MI) Regimen (N=74) | Cyclosporin Regimen (N=71)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 0 | 0 | 0
Fructose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 0 | 0 | 0
Urinary fistula (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Zygomycosis (Infections and infestations) | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 1
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 1 | 0
Cytomegalovirus enteritis (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1
Infective myositis (Infections and infestations) | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1 | 0
Prostatic dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 2 | 1 | 3
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 8 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 3 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Lymphocele (Vascular disorders) | 2 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 4 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0
Graft loss (Injury, poisoning and procedural complications) | 0 | 1 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0
Meningorrhagia (Nervous system disorders) | 0 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 3 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 2 | 1
Salivary gland disorder (Gastrointestinal disorders) | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0
Arterial stenosis (Vascular disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
BK virus infection (Infections and infestations) | 1 | 0 | 0
Cyst rupture (General disorders) | 0 | 0 | 0
Cytomegalovirus gastroenteritis (Infections and infestations) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 8 | 4 | 6
Renal cyst infection (Infections and infestations) | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0
Transplant rejection (Immune system disorders) | 20 | 18 | 9
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 4
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 4 | 5 | 7
Depression (Psychiatric disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 3
Endophthalmitis (Infections and infestations) | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 2
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0
Kidney transplant rejection (Immune system disorders) | 3 | 2 | 2
Localised infection (Infections and infestations) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 2 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 2 | 2 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0
Urinoma (Renal and urinary disorders) | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Vesical fistula (Renal and urinary disorders) | 1 | 1 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Catheter removal (Surgical and medical procedures) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Ureteral necrosis (Renal and urinary disorders) | 1 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Blood creatinine abnormal (Investigations) | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cavernous sinus thrombosis (Infections and infestations) | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Fat necrosis (General disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0
Fungal test positive (Investigations) | 0 | 0 | 0
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Quadriplegia (Nervous system disorders) | 0 | 0 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept: Less-intensive (LI) Regimen (N=71) | Belatacept: More-intensive (MI) Regimen (N=74) | Cyclosporin Regimen (N=71)
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 4 | 0
Chest pain (General disorders) | 3 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 | 9 | 7
Hypotension (Vascular disorders) | 4 | 5 | 4
Leukopenia (Blood and lymphatic system disorders) | 13 | 13 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4
Pain (General disorders) | 5 | 7 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5 | 2
Tremor (Nervous system disorders) | 10 | 8 | 14
Abdominal distension (Gastrointestinal disorders) | 4 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 6
Acne (Skin and subcutaneous tissue disorders) | 4 | 6 | 2
Fatigue (General disorders) | 6 | 6 | 9
Headache (Nervous system disorders) | 10 | 13 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 3 | 7
Insomnia (Psychiatric disorders) | 19 | 12 | 17
Oral candidiasis (Infections and infestations) | 2 | 4 | 4
Tachycardia (Cardiac disorders) | 4 | 4 | 5
Blood creatinine increased (Investigations) | 8 | 7 | 11
Bronchitis (Infections and infestations) | 7 | 4 | 2
Flatulence (Gastrointestinal disorders) | 4 | 3 | 2
Graft dysfunction (Injury, poisoning and procedural complications) | 9 | 7 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 4 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 5 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 6 | 4
Abdominal pain lower (Gastrointestinal disorders) | 4 | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 6
Dysuria (Renal and urinary disorders) | 3 | 4 | 1
Generalised oedema (General disorders) | 3 | 6 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 24 | 14 | 15
Nasopharyngitis (Infections and infestations) | 10 | 11 | 12
Nausea (Gastrointestinal disorders) | 18 | 19 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 6
Proteinuria (Renal and urinary disorders) | 6 | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 12 | 13 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 9 | 4
Constipation (Gastrointestinal disorders) | 22 | 16 | 17
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Oedema peripheral (General disorders) | 20 | 23 | 22
Pyrexia (General disorders) | 12 | 12 | 11
Rash (Skin and subcutaneous tissue disorders) | 2 | 7 | 6
Transplant rejection (Immune system disorders) | 5 | 3 | 4
Urinary tract infection (Infections and infestations) | 18 | 17 | 19
Urine output decreased (Investigations) | 2 | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 6
Acidosis (Metabolism and nutrition disorders) | 1 | 3 | 6
Cytomegalovirus infection (Infections and infestations) | 7 | 9 | 10
Depression (Psychiatric disorders) | 3 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 19 | 17 | 16
Dyspepsia (Gastrointestinal disorders) | 6 | 7 | 3
Haematuria (Renal and urinary disorders) | 5 | 5 | 6
Hirsutism (Skin and subcutaneous tissue disorders) | 3 | 1 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 6 | 9
Hypertension (Vascular disorders) | 17 | 16 | 19
Metabolic acidosis (Metabolism and nutrition disorders) | 4 | 2 | 1
Oedema (General disorders) | 8 | 6 | 10
Procedural pain (Injury, poisoning and procedural complications) | 17 | 14 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 5
Dizziness (Nervous system disorders) | 3 | 4 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Incision site pain (Injury, poisoning and procedural complications) | 16 | 15 | 9
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 6
Chills (General disorders) | 5 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 3 | 6
Leukocytosis (Blood and lymphatic system disorders) | 4 | 2 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 5
Vomiting (Gastrointestinal disorders) | 14 | 10 | 8
White blood cell count decreased (Investigations) | 1 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.